CLINICAL TRIAL: NCT05021289
Title: Effect of the Practice of Guided Imagery on the Perceived Stress Level in High-Risk Pregnancies: Randomized Single-Blind Trial
Brief Title: Guided Imagery on the Perceived Stress Level in High-Risk Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nursel Alp Dal (Other)
Responsible Party: Sponsor-Investigator, Nursel Alp Dal, Assistant Professor, Munzur University
Organization: Munzur University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MunzurUn
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: High Risk Pregnancy
Keywords: Guided Imagery; Perceived Stress Level; High-Risk Pregnancies.
MeSH Terms: interventions — Imagery, Psychotherapy

STUDY DESIGN:
Intervention Model Description: Designed as a prospective randomized single-blind trial, the research was performed with the participation of a total of 128 women who had high-risk pregnancies and received inpatient treatment on 1 February - 1 May 2021 at the perinatology service of a maternity and children's hospital located in the Anatolian side of Istanbul province of Turkey (64 pregnant women in the experimental group, 64 pregnant women in the control group).
Who Masked: Participant
Masking Description: care provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided İmagery (Experimental): • participants were given one session of guided imagery.
  Interventions: Behavioral: guided imagery
- control group (No Intervention): No intervention was applied on the control group patients.

INTERVENTIONS:
Behavioral: guided imagery — guided imagery
  Arms: Guided İmagery

SUMMARY:
This research was conducted to identify the effect of the practice of Guided Imagery on the perceived stress level in high-risk pregnancies.

DETAILED DESCRIPTION:
Designed as a prospective randomized single-blind trial, the research was performed with the participation of a total of 128 women who had high-risk pregnancies and received inpatient treatment on 1 February - 1 May 2021 at the perinatology service of a maternity and children's hospital located in the Anatolian side of Istanbul province of Turkey (64 pregnant women in the experimental group, 64 pregnant women in the control group).

ELIGIBILITY:
Inclusion Criteria:• Having a high-risk pregnancy

* Being aged 18 years or above
* Agreeing to participate in the study
* Being literate in Turkish

Exclusion Criteria:

* The pregnant women who voluntarily wanted to leave the research at any stage after being included in the study, could not communicate verbally, had a visual or hearing disorder, and were previously diagnosed with a psychiatric disease were excluded from the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The research population was comprised of all women who had high-risk pregnancies and received treatment at the perinatology service of the aforementioned hospital in the above period
Enrollment: 128 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale. | • The first practice of guided imagery was performed face-to-face with pregnant women. At the end of 20 minutes, the pregnant women's stress levels were reevaluated by using the Perceived Stress Scale.
  Evaluation of the stress level of pregnant women with the Perceived Stress Scale. Comprised of 14 items in total, the scale was designed to measure the extent to which circumstances in one's life are perceived as stressful. The respondents evaluate the items based on a five-point Likert scale that is scored from '0: Never' to '4: Very Often'. Seven positively-stated items are reverse scored. The minimum and maximum scores to be obtained from the scale are successively 0 and 56 points. A high score obtained from the scale indicates that the respondent has high-level stress perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Munzur University, Tunceli, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No